CLINICAL TRIAL: NCT00572741
Title: Treating Oxidative Stress and the Metabolic Pathology of Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 59538; 59538
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Autistic Disorder
Keywords: Autism; vitamin B 12; glutathione
MeSH Terms: conditions — Autistic Disorder | interventions — Vitamin B 12; Folic Acid; Hydroquinones; Ascorbic Acid; Cod Liver Oil; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nutritional supplementation
  Interventions: Dietary Supplement: B12; Dietary Supplement: folate; Dietary Supplement: B complex; Dietary Supplement: vitamin C; Dietary Supplement: cod liver oil; Dietary Supplement: Mineral complex; Dietary Supplement: carnitine
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B12 — Methylcobalamin Dose: 75 μg/kg every 3 days
  Arms: 1
Dietary Supplement: Placebo — cellulose
  Arms: 2
Dietary Supplement: folate — Folinic acid: Dose: 400 µg twice a day (BID)
  Arms: 1
Dietary Supplement: B complex — B-Complex: B-1 (3 mg); B-2 (3.4 mg); B-352 (20 mg); B-6 (4 mg;) Pantothenic Acid(10 mg); Biotin (300 mcg); pyridoxal (25mg)
  Arms: 1
Dietary Supplement: vitamin C — Vitamin C 500 mg
  Arms: 1
Dietary Supplement: cod liver oil — Cod liver oil 1/2 teaspoon
  Arms: 1
Dietary Supplement: Mineral complex — Magnesium citrate (200 mg); Selenium (50 mcg); Zinc picolinate (25 mg); Molybdenum (50 mcg); Calcium citrate (400 mg)
  Arms: 1
Dietary Supplement: carnitine — Acetyl L-Carnitine Dose: 250 mg
  Arms: 1

SUMMARY:
Hypothesis: Many children with autism have impaired methylation and antioxidant/detoxification capacity and chronic oxidative stress. A targeted nutritional intervention that is designed to correct the metabolic imbalance will normalize their metabolic profile and improve measures of autistic behavior.

DETAILED DESCRIPTION:
Hypothesis and Specific Aims Hypothesis: A significant proportion of autistic children have impaired methylation and antioxidant/detoxification capacity resulting in chronic oxidative stress. Targeted nutritional intervention that is designed to correct the metabolic imbalance will significantly improve their metabolic profile and improve measures of autistic behavior.

If proven correct, this hypothesis could generate specific biomarkers to define individual behavioral phenotypes within the autism spectrum and indicate targeted treatment options to reduce and possibly prevent the clinical and behavioral manifestations of autism.

Specific Aim 1. To screen children with a diagnosis of autism for evidence of impaired methylation (↓SAM/SAH) and impaired antioxidant capacity (↓GSH/GSSG)

Specific Aim 2. Children who exhibit evidence of impaired methylation and antioxidant capacity will be randomized into a double blind placebo-controlled parallel group trial of targeted nutritional intervention designed to correct metabolic deficiencies and imbalance and to improve scores on standardized behavioral evaluation tests.

The two specific aims (Study Phase 1 and 2 respectively) are designed to increase the understanding of the metabolic factors that contribute to development and clinical manifestations of autism. We anticipate that the knowledge gained from the successful achievement of our aims will provide an important new metabolic dimension to early diagnosis and clinical management of autistic children.

Rationale:

Although the efficacy of nutritional intervention in autistic children has been evaluated in numerous reports in the literature, these studies are generally considered inconclusive. Despite positive results, most have been criticized for small sample size, poor study design, lack of placebo group, heterogeneity of diagnosis, and/or efficacy based on subjective parent report. Because of these limitations, none of the studies have successfully demonstrated that targeted nutritional supplementation can be an efficacious treatment approach for autistic children. Consequently, there is a real need for large well-designed placebo-controlled studies with intervention strategies based on metabolic or nutritional endpoints that can be followed for treatment efficacy and related to quantitative improvements in standardized behavioral testing conducted in a blinded manner.

While knowledge of individual nutrient response efficacy is a desirable goal, the reality is that all metabolic pathways are inextricably interwoven and interdependent such that perturbation of one pathway will inevitably affect other pathways. This means that addressing a deficit in one single pathway is highly likely to alter requirements and possibly negatively affect other interdependent pathways. A broad spectrum balanced approach to correct the observed metabolic imbalance in autistic children is the basis for the intervention strategy proposed in the present intervention trial.

Because the efficacy for nutritional intervention in autistic children is based solely on anecdotal evidence, a placebo-controlled double blind study is now clearly needed to establish scientifically in a carefully designed clinical trial whether this approach has efficacy or whether it does not. Either outcome will provide valuable information to parents and physicians currently recommending these supplements. If the outcome indicates therapeutic efficacy, this information will be published in the scientific literature so that mainstream medicine is aware of this approach. If the outcome indicates a lack of efficacy, dissemination of this information will be important to prevent needless wasting of monetary resources.

Targeted Metabolic Therapy Abnormalities in folate, methionine and glutathione metabolism will directly or indirectly affect phospholipid metabolism, mitochondrial energy metabolism, detoxification/antioxidant capacity, and mineral cofactor availability. Therefore, correction of an imbalance in folate/methionine and glutathione metabolism requires a global and targeted nutritional intervention strategy rather than isolated single nutrient supplementation. A nutritionally balanced diet consisting of fruits, vegetables and meat will be encouraged. Although helpful, a diet-only approach is generally considered to be insufficient to overcome genetically-based chronic metabolic imbalance. Further, control over nutrient intake between individual children is impossible with diet-only intervention and may be complicated by sensory issues and restricted dietary preferences in autistic children. Therefore, we have designed a balanced and targeted supplementation strategy specifically designed to support and correct observed metabolic imbalances in autistic children.

Based on these considerations and extensive literature review, the supplements have been selected to impact three core cellular functions that may be impaired with chronic oxidative stress in many children with autism:

1. Decreased SAM/SAH ratio and cellular methylation capacity: the methionine synthase reaction and SAM synthesis are redox sensitive and inactivated by low GSH and oxidative stress. 40-43
2. Cell membrane integrity: membrane lipid peroxidation occurs with oxidative stress as evidenced by elevated isoprostanes in autistic children.24,44,45
3. Antioxidant and detoxification support (mitochondrial and cytosolic): Glutathione levels and redox ratio are significantly reduced in many autistic children.1,42,46

The selection of supplements and dose level was made in consultation with Bryan Jepson MD, who recently published a book entitled "Changing the course of autism: a scientific approach for parents and physicians" (available to IRB upon request). Dr. Jepson is a parent of an autistic child and a physician who has treated hundreds of autistic children in his autism practice in Austin, Texas. The supplements are highly unlikely to produce toxic side effects based on previous published studies in the scientific literature showing efficacy in children without toxic side effects. We have created a table (submitted and approved by the IRB) indicating that for each micronutrient, the supplement level falls below the IOM designated safe upper limit. The table also allows a comparison of the safe upper limit with the study dose for each of the micronutrients and provides quotes from the scientific literature indicating that intakes above our supplement levels have been shown to be non-toxic. Stephen Kahler MD, clinical geneticist and member of our research team, and our PCP consultant, Bryan Jepson MD, both agree that these levels are safe and likely to be efficacious. Indeed, the same supplement levels are commonly prescribed by PCPs who are currently treating thousands of autistic children without report of toxic side effects. Finally, we consulted locally with Donald Mock, MD PhD, who also expressed confidence in the safety of the recommended supplements and dose levels.

The selected supplements are all available over-the counter (OTC) and considered by the FDA to be GRAS (generally recognized as safe) and fall under safety regulations of the DSHEA Act (Dietary Supplement Health and Education Act). We have chosen to obtain the supplements from a highly reputable compounding pharmacy, Kirkman Laboratories to avoid additives and food dyes often present in OTC supplements that may cause negative side effects in some autistic children. Kirkman Laboratories has been manufacturing prescription drugs and nutritional supplements since 1949 using Standard Operating Procedures required by the FDA (FDA registration 3025062). Their manufacturing process is based on "Good Manufacturing Practices" as defined by the FDA and is monitored by an independent quality control department.

Our research team is strengthened by the continued participation of the ACH Research Pharmacist, who has been working closely with Kirkman Laboratories. The ACH Research Pharmacist will receive and distribute the supplements/placebos and will assure proper storage conditions as he has for our open label study, Protocol #28839.

Behavioral Tests:

Each of the tests was chosen based on the recommendation of our consultant and certified behavioral analyst, Doreen Granpesheh PhD. These tests are deemed most likely to detect change with treatment intervention and when appropriate (e.g., ADOS) will be administered by ACH Pediatric Psychologists. The ADOS behavior test will be videotaped. A second behavior analyst will evaluate a random set of these video recordings to confirm inter-rater reliability.

Autism Diagnostic Observation Schedule (ADOS) is the "gold standard" for assessing and diagnosing autism and pervasive developmental disorder (PDD) across ages, developmental levels, and language skills.

Vineland Adaptive Behavior Scales (VABS) provides an age-adjusted overall autism severity score and individual scores for regressive/expressive verbal and non-verbal communication, fine and gross motor skills, and interpersonal behavior.

The Social Responsiveness Scale (SRS) distinguishes autism spectrum conditions from other child psychiatric conditions by identifying presence and extent of autistic social impairment .Completed by a parent the SRS provides a clear picture of a child's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance and autistic preoccupations and traits.

Preschool Language Scale Fourth Edition (PLS-4) is a standardized test of auditory comprehension and expressive communication for infants and toddlers. The auditory comprehension subscale assesses basic vocabulary, concepts and grammatical markers in preschool and higher-level abilities such as complex sentences, making comparisons and inferences in older children. The expressive communication subscale asks preschoolers to name objects, use concepts that describe objects, express quantity, use grammatical markers, etc. It also includes word segmentation, completing analogies, and telling a short story in sequence.

The Clinical Global Impression (CGI) is a tool used to pick up subtle behavior changes that may not be caught by the other behavior tests. The CGI is 3 item observer rated scale that measures illness severity, global improvement or change, and therapeutic response. This tool is widely available to be used in the public domain. For our study, the Pediatric Psychologists will be using the illness severity and global improvement sections of this tool.

The Block Food Frequency Questionnaire, the Child's Sleep Habits Questionnaire, the GI Symptom Inventory, the Pediatric Quality of Life Questionnaire (PQOL), and the Parental Stress Index (PSI) are completed by the parent(s) with the assistance of the study nurse.

Supplement Doses, Formulation and Administration Targeted metabolic support is based on metabolic evidence of oxidative stress and/or impaired methylation capacity. The supplements will be in the form of methyl B12 pre-loaded syringes (previously approved by UAMS IRB [protocol #28839] and the FDA [IND # 71459]), small capsules (folinic acid and carnitine), powder (minerals and antioxidants), and a liquid (cod liver oil and essential fatty acids). The placebos (cellulose) will be prepared in identical form by Kirkman Laboratories. The Methyl B12 pre-loaded syringes and placebos will be prepared in identical form by Custom Compounding Pharmacy

The rationale and dosing schedule for each supplement is based on its established efficacy in the following categories:

1. For SAM/SAH and methylation capacity:

   Injectible methylB12; Folinic acid.
2. Mineral cofactors for enzymes involved in methylation and transsulfuration:

   Magnesium citrate47,48 ; Selenium 49,51, Zinc picolinate50,51, Molybdenum51; Calcium citrate51; Vitamin D 52.
3. For Antioxidant and detoxification support (cytosolic and mitochondrial):

   Multivitamin powder containing: Vitamin C 52; Vitamin E 52,53; Vitamin K 52 ; B-Complex 52: B-1; B-2 52; B-3 52; B-6 52, Pantothenic Acid 52; Biotin 52; pyridoxal 52, Taurine 54 ; Pycnogenol 55,56,57; CoQ 10 58; Choline 52.
4. For Membrane integrity: Cod Liver Oil plus essential fatty acids 53, Acetyl L-Carnitine 59,60

ELIGIBILITY:
Inclusion Criteria:

* ADOS and DSM-IV (299.0) diagnosis of Autistic Disorder
* Both sexes
* Age range 3-7

Exclusion Criteria:

* Pervasive Developmental Disorder, Not Otherwise Specified (PDD-NOS)
* Asperger's
* Rett syndrome
* Fragile X
* Tuberous sclerosis or other genetic conditions associated with autism
* Frequent seizures
* Recurrent or current infection
* Severe gastrointestinal distress
* Recent supplement use

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Behavioral test scores | 4 months

SECONDARY OUTCOMES:
Plasma metabolic profile | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jill James, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Background] James SJ, Melnyk S, Jernigan S, Cleves MA, Halsted CH, Wong DH, Cutler P, Bock K, Boris M, Bradstreet JJ, Baker SM, Gaylor DW. Metabolic endophenotype and related genotypes are associated with oxidative stress in children with autism. Am J Med Genet B Neuropsychiatr Genet. 2006 Dec 5;141B(8):947-56. doi: 10.1002/ajmg.b.30366. PMID 16917939
- [Result] James SJ, Melnyk S, Fuchs G, Reid T, Jernigan S, Pavliv O, Hubanks A, Gaylor DW. Efficacy of methylcobalamin and folinic acid treatment on glutathione redox status in children with autism. Am J Clin Nutr. 2009 Jan;89(1):425-30. doi: 10.3945/ajcn.2008.26615. Epub 2008 Dec 3. PMID 19056591